CLINICAL TRIAL: NCT00191074
Title: Phase III Study of Humatrope in Non-Growth Hormone Deficient Children With Short Stature
Brief Title: Amendment (g) Unblinded Extension Phase of Somatropin in Patients With Idiopathic Short Stature
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 843; B9R-MC-GDCH
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-03-09 (Estimated); Status verified 2007-03

CONDITIONS: Growth Disorder
MeSH Terms: conditions — Growth Disorders | interventions — Human Growth Hormone; WW Domain-Containing Oxidoreductase

INTERVENTIONS:
Drug: somatropin, rDNA origin, for injection

SUMMARY:
After approval of amendment (g), patients who were still receiving study drug at the time were scheduled for a study visit. In addition, patients who had discontinued early from the core, blinded phase of the study were contacted.

All of these patients were offered the opportunity to enter the unblinded extension phase (if they met eligibility criteria) and continue somatropin treatment (regardless of initial treatment randomization) until they reached final height.

ELIGIBILITY:
Inclusion Criteria:

Participation in core, blinded phase and ability to be contacted by investigators.

For patients who were on treatment at the time of amendment (g), growth velocity greater than or equal to 1.5 cm/year measured over the prior 12-month period. For patients who had chosen to discontinue treatment in the core, blinded phase, bone age less than or equal to 16 years for boys and less than or equal to 14 years for girls.

Exclusion Criteria:

Diabetes mellitus.

History, evidence or signs of active malignancy within 5 years prior to the start of the extension phase.

Any condition or medication that, in the opinion of the investigators, might significantly increase the risk or decrease the efficacy of growth hormone therapy.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11
Dates: Start 2001-02; Study Completion 2006-01

PRIMARY OUTCOMES:
Every 6 months: physical exam, pubertal staging, height, weight, and adverse event collection.
Every year: arm span measurements, head circumference measurements, x-ray for bone age, and
laboratory blood draws.

SECONDARY OUTCOMES:
Not applicable for Amendment (g).

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethesda, Maryland, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com